CLINICAL TRIAL: NCT00987064
Title: Clinical Effects of Purified Air Administered to the Breathing Zone in Allergic Asthma
Brief Title: Clinical Effects of Temperature Controlled Laminar Airflow (TLA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Airsonett AB (Industry)
Collaborators: Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Quintiles, Inc. (Industry)
Responsible Party: Prof. Dr. Gunilla Hedlin, Head of Activity, Karolinska Universitety hospital Solna Sweden
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Air 3-01
Record Dates: First submitted 2009-09-28; First posted 2009-09-30 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2009-09

CONDITIONS: Asthma; Perennial Allergy
Keywords: Protexo; Asthma; Temperature controlled Laminar Airflow; Perennial allergy; Quality of life; MiniAQLQ; FeNO; FEV1; PEF
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temperature controlled Laminar Airflow (Active Comparator): Active treatment with Temperature controlled Laminar Airflow (TLA)
  Interventions: Device: Temperature controlled Laminar Airflow (Protexo)
- Placebo TLA (Placebo Comparator): Placebo treatment with TLA (no filtration function)
  Interventions: Device: Placebo TLA

INTERVENTIONS:
Device: Temperature controlled Laminar Airflow (Protexo) — The intervention is designed to reduce the allergen load in the patients breathing zone by vertically displacing the allergens, originating from the bed and the ambient room environment, with a temperature controlled laminar airflow (TLA) during night sleep. The airflow is filtered through a high efficiency particulate air filter(HEPA), slightly cooled and ''showered'' over the subject. Due to the higher density, the cooled air descends slowly, and displaces the allergens from the breathing zone.
  Other Names: Protexo
  Arms: Temperature controlled Laminar Airflow
Device: Placebo TLA — TLA treatment with disabled filtration function
  Arms: Placebo TLA

SUMMARY:
The purpose of this study is to determine whether clean air administered to the breathing zone with Temperature controlled Laminar Airflow (TLA) during night is effective in the treatment of perennial allergic asthma.

DETAILED DESCRIPTION:
Background: Exposure to inhaled allergens is a pathogenetic factor in allergic asthma. However, most studies that previously looked at air cleaning devices have shown little or no effect on patients with perennial allergic asthma. Aims and objectives: This study aims to investigate a novel treatment, TLA, using temperature controlled laminar airflow with a very low particle concentration directed to the breathing zone of teenagers and adults with allergic asthma during night sleep. The hypothesis is that the decreased allergen exposure during the night will have an effect on bronchial inflammation and quality of life. Method: Patients are randomized to start with active or placebo treatment for 10 weeks. All patients receive both active and placebo treatment with unfiltered air, with a 2-week wash-out period in between treatments. Maintenance treatment with inhaled corticosteroids is unaltered during the trial period. Health related quality of life (miniAQLQ)is the primary effectiveness measure. Exhaled nitric oxide (FeNO) and spirometry are also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed for asthma for more than 1 year.
* More than 12% reactivity in FEV1 on bronchodilating medication or less than 90% of the FEV1 reference value according to Hedenström.
* Perennial allergy
* At least 3-mm wheal reaction in a skin prick test to at least one of following: House dust, Mold spores, dust mites, animal hair and dander.
* Little or no reactivity to other inhalant allergens.
* No known allergy to another inhalant allergen or chemical to which there is exposure in winter time.
* No allergen injection treatment in the preceding 2 years.
* A history of a requirement for daily medication for asthma including;

  * 400µg steroid medication (Pulmicort or equal) for children and 800µg for adults.
  * Beta agonist treatment on less than 4 days per week.
* Willingness to follow the clinical trial protocol, including medications, baseline and follow-up visits and procedures.

Exclusion Criteria:

* Inclusion in another Allergen avoidance program.
* Smoking in the family
* Participation in a drug trial

Ages: 12 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed by mini Asthma Quality of Life Questionnaire (miniAQLQ) | Every 2 weeks of the study period

SECONDARY OUTCOMES:
Airway inflammation measurement assessed by Exhaled nitric oxide (FeNO) | Every 5 week of the study period
Lung function (FeV1, PEF) | Every 5 week of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Pedroletti, MD, PhD., Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - University Hospital, Linkoeping, Linköping
  - Karolinska University Hospital, Stockholm

REFERENCES:
- [Background] Pedroletti C, Millinger E, Dahlen B, Soderman P, Zetterstrom O. Clinical effects of purified air administered to the breathing zone in allergic asthma: A double-blind randomized cross-over trial. Respir Med. 2009 Sep;103(9):1313-9. doi: 10.1016/j.rmed.2009.03.020. Epub 2009 May 13. PMID 19443189